CLINICAL TRIAL: NCT05379166
Title: Phase II Study of Clinical Efficacy of Venetoclax in Combination With Azacitidine in Patients With Therapy Related Myelodysplastic Syndrome (t-MDS)
Brief Title: Venetoclax and Azacitidine for Treatment of Therapy Related or Secondary Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uma Borate (Other)
Responsible Party: Sponsor-Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20420; NCI-2021-08484 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-03-15; First posted 2022-05-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Secondary Myelodysplastic Syndrome; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, azacitidine) (Experimental): Patients receive venetoclax PO QD on days 1-14 and azacitidine IV over 10-40 minutes on days 1-7 or days 1-5 of week 1 and days 1 and 2 of week 2. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies the effect of venetoclax and azacitidine in treating patients with therapy related or secondary myelodysplastic syndrome. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax in combination with azacitidine may work better in treating patients with therapy related or secondary myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the proportion of participants that achieve a complete remission following treatment with azacitidine and venetoclax.

SECONDARY OBJECTIVES:

I. Assess safety of azacitidine and venetoclax combination therapy. II. Determine the overall response rate (ORR). III. Determine the complete cytogenetic response rate (CCyR). IV. Determine the duration of response (DOR). V. Estimate event-free survival (EFS). VI. Estimate overall survival (OS). VII. Determine combined hematologic improvement rate (HIR). VIII. Determine red blood cell transfusion independence rate. IX. Determine platelet transfusion independence rate. X. Determine proportion of participants whose disease transforms to acute myeloid leukemia (AML).

XI. Determine proportion of participants that proceed to allogeneic hematopoietic stem cell transplantation (alloHSCT).

XII. Compare response criteria between the 2006 International Working Group (IWG) and 2023 IWG criteria.

EXPLORATORY OBJECTIVES:

I. Determine baseline frequencies of cytogenetic aberrations and their relationships to response to study therapy.

II. Estimate progression-free survival (PFS). III. Obtain quality of life (QoL) information from patient-reported responses to Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 7a and European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) - Core 30 (C30) questionnaires.

OUTLINE:

Patients receive venetoclax orally (PO) once daily (QD) on days 1-14 and azacitidine intravenously (IV) over 10-40 minutes on days 1-7 or days 1-5 of week 1 and days 1 and 2 of week 2. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 6 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Age >= 18 years at time of informed consent. Both men and women and members of all races and ethnic groups will be included
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Previously untreated therapy related myelodysplastic syndrome (t-MDS) with Revised International Prognostic Scoring System (IPSS-R) risk categories Intermediate, High or Very High (i.e., minimum IPSS-R score of 3.5) and presence of < 20% bone marrow blasts per bone marrow biopsy/aspirate
* Patients with t-MDS which is defined as patients who have had prior anti-cancer therapy including chemotherapy and/or radiation therapy
* Aspartate aminotransferase (AST) < 3.0 x upper limit of normal (ULN) x upper limit of normal (ULN; local laboratory)
* Alanine aminotransferase (ALT) < 3.0 x ULN x ULN
* Total bilirubin =< 2 x ULN (except for patients with known Gilbert's syndrome)
* Creatinine clearance >= 30 mL/min OR serum creatinine < 1.5 x the ULN
* White blood cell (WBC) count =< 10,000/uL

  * Note: Treatment with hydroxyurea is permitted to lower the WBC to reach this inclusion criterion. The WBC should be determined >= 24 hours after the last dose of hydroxyurea. The last dose of hydroxyurea should not be administered =< 3 days prior to the first dose of azacitidine
* Females of childbearing potential (FOCBP) must agree to adequate contraception (1 form of contraception or abstinence) from the screening visit until 30 days following the last dose of venetoclax. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately

  * FOCBP are those who have not been surgically sterilized or have not been free from menses for > 1 year without an alternative medical cause
* Male patients of childbearing potential having intercourse with females of childbearing potential must agree to abstain from heterosexual intercourse or have their partner use 2 forms of contraception from the screening visit until 90 days after the last dose of study treatment. They must also refrain from sperm donation from the screening visit until 90 days following the last dose of study treatment

Exclusion Criteria:

* Participant has received prior therapy with a venetoclax or other BH3 mimetic. Note: Prior supportive care in form of transfusions or growth factors, etc., is not considered prior therapy. Supportive care should be discontinued >= 14 days prior to the first dose of study drug. Subjects may continue oral corticosteroids for management of conditions other than MDS (e.g., asthma, rheumatoid arthritis) at a stable daily dose equivalent to =< 10 mg prednisone during screening and study participation
* Subject has a diagnosis other than previously untreated de novo MDS with IPSS-R risk categories Intermediate, High or Very High, including:

  * MDS with IPSS-R risk categories Very Low or Low (overall IPSS score < 3)
  * MDS evolving from a pre-existing myeloproliferative neoplasm (MPN)
  * MDS/MPN including chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (CML), juvenile myelomonocytic leukemia (JMML) and unclassifiable MDS/MPN
* Patients who are suitable for and willing to receive intensive chemotherapy or eligible to proceed to allogeneic stem cell transplantation without additional therapy
* Known history of testing positive for Human Immunodeficiency Virus (HIV) infections, Hepatitis B, or Hepatitis C. For countries where HIV status is mandatory: testing positive for HIV during screening using a local test.
* Clinically significant ventricular arrhythmia (e.g., ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure
* Patients with uncontrolled infection will not be enrolled until infection is treated and under control
* Hypersensitivity to any study agent when administered alone. Any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol
* Any psychiatric illness that prevents patient from informed consent process
* Pregnant of breastfeeding at the time of enrollment
* Subject has received allogeneic HSCT or solid organ transplantation
* Subject has a concurrent active malignancy requiring treatment or with an expected life expectancy less than 1 year with the exception of below. Any subject with a concurrent active malignancy will be reviewed by the PI for eligibility prior to enrollment

  * Adequately treated in situ carcinoma of the cervix uteri
  * Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin
  * Asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy
* Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Ongoing systemic infection (viral, bacterial, or fungal)
  * Acute pneumonia
  * Febrile neutropenia
* Subject has received strong or moderate CYP3A inducers within 7 days prior to the first dose of study drug
* Subject has received strong or moderate CYP3A inhibitors within 7 days prior to the first dose of study drug
* Subject has consumed one or more of the following within 3 days prior to the first dose of study drug:

  * Grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * Star fruit (carambola)
* Subject has a malabsorption syndrome or other condition that precludes an enteral route of administration
* Subject has history of a cardiovascular, endocrinologic, hepatic, immunologic metabolic, neurologic, psychiatric, pulmonary, renal disease, or any other condition that in the opinion of the investigator would adversely affect his/her participation in this study or interpretation of study results
* Subject has received a live attenuated vaccine within 4 weeks prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) | At the end of Cycle 4 (each cycle is 28 days) or earlier based on bone marrow results
  Defined by 2023 International Working Group (IWG) criteria. A point estimate and 95% exact (i.e., Clopper-Pearson) confidence interval will be computed for the CR rate within the efficacy-evaluable population.

SECONDARY OUTCOMES:
Treatment emergent adverse events (AEs) | Up to 30 days after last dose of study drug
  AEs defined by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Participant-level tallies of treatment emergent adverse events will be reported overall and by System Organ Class (according to Medical Dictionary for Regulatory Activities [MedDRA]), with separate tables of frequency counts and percentages made for grade >= 3 AEs and serious AEs. Moreover, AE attributions will be utilized so that specific categories of study drug-related adverse reactions (e.g., at least possibly related; definitely related) can also be tallied and summarized by Organ Class.
Overall response rate (ORR) | At the end of the last cycle of study drug (each cycle is 28 days)
  The ORR rate (proportion of participants achieving a CR, CR equivalent, partial remission [PR], CR with limited count recovery (CRL), CR with partial hematologic recovery (CRh), or Hematologic Improvement (HI)) will be described with a point estimate and 95% exact confidence interval for the efficacy-evaluable population.
Cytogenetic response rate (CCyR) | At the end of the last cycle of study drug (each cycle is 28 days)
  The CCyR rate, applied to the set of participants whose bone marrow shows an abnormal karyotype at baseline and who are subjected to at least one post- study drug chromosomal G banding analysis, will be estimated along with a 95% exact confidence interval.
Overall survival (OS) | From date of death or the last known alive date for participants who withdraw from or complete the study without dying, assessed up to 24 months
  OS distributions will be estimated with the Kaplan Meier method, with estimates for median survival and survival rates at landmark times (e.g., 1-year) provided.
Duration of response (DOR) | From earliest occurrence of PR, mCR, or CR to onset of progressive disease, assessed up to 24 months
Event free survival (EFS) | From event date or date of last clinic visit for participants without an event during the study period, assessed up to 24 months
  EFS distributions will be estimated with the Kaplan Meier method, with estimates for median survival and survival rates at landmark times (e.g., 1-year) provided.
Hematologic improvement rate (HIR) | At the end of the last cycle of study drug (each cycle is 28 days)
  Within the hematologic improvement analysis set, the number and percentage (with exact 95% confidence interval) of participants with HIR will be listed.
Rates of hematologic improvement-erythrocytes (HI-E) | At the end of the last cycle of study drug (each cycle is 28 days)
  Rates of HI-E will be computed along with exact 95% confidence intervals and associated sample sizes.
Rates of hematologic improvement-platelets (HI-P) | At the end of the last cycle of study drug (each cycle is 28 days)
  Rates of HI-P will be computed along with exact 95% confidence intervals and associated sample sizes.
Rates of hematologic improvement-neutrophils (HI-N) | At the end of the last cycle of study drug (each cycle is 28 days)
  Rates of HI-N will be computed along with exact 95% confidence intervals and associated sample sizes.
Percentage of participants who have disease that transforms to acute myeloid leukemia (AML) | End of study follow-up period (24 months after last dose of study drug)
  Will be estimated with exact 95% confidence intervals for the intent to treat (ITT) population, safety, and efficacy populations.
Percentage of participants who proceed to allogeneic hematopoietic stem cell transplantation | 12 months after last dose of study drug
  Will be estimated with exact 95% confidence intervals for the ITT population, safety, and efficacy populations.
Percentage of patients achieving CR, CR equivalent, CRi, CRh, PR, or HI | From first dose of study drug to end of last cycle of study drug (each cycle is 28 days)

OTHER OUTCOMES:
Detection of cytogenetic abnormalities | Up to 12 months or last bone marrow exam
  Detection of cytogenetic abnormalities (e.g., all or partial deletions of chromosome 5 or 7) will be summarized for baseline and, if available, post-treatment karyotype results with point and 95% exact confidence interval estimates for (i) all participants and (i) within specific response groups (e.g., CR). Fisher's exact test will be utilized to determine the association between the baseline occurrence of each common chromosomal abnormality and ORR group (i.e., "overall" responders with a best response of PR, mCR, or CR versus [vs.] non-responders with stable disease [SD] or partial disease [PD]).
Biometric measures recorded by the FitBit (e.g., heart rate, number of steps taken, activity time, calories burned) | At the end of cycle 1 of study drug (each cycle is 28 days)
  Biometric measures (heart rate, number of steps, distance, minutes of activity, number of calories burned) from participants agreeing to wear a FitBit device will be summarized descriptively (median, interquartile range [IQR], mean, standard deviation [SD], range) for day and week increments and correlated with (i) Eastern Cooperative Oncology Group (ECOG) performance status using the Kruskal-Wallis test and (ii) physical function assessment results such as grip strength and gait speed using correlation coefficients. The FitBit measures of activity will also be analyzed for time trends and their averages compared with clinical outcomes (e.g., best response, hematologic improvement, number of cycles of study drug).
Patient-reported outcomes (PROs) | Up to 12 months or end of treatment clinical visit
  Patient-reported outcomes from Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue SF 7a and European Organisation for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) - Core 30 (C30) questionnaires will be collected at baseline (within 3 days of commencing study drug on cycle 1, day 1) and pre-dosing on day 1 of cycles 2, 3, 5, 7, and every third subsequent cycle through the end of treatment visit. These PROs will be quantified using the respective questionnaire's scoring manual.

CONTACTS AND LOCATIONS:
Overall Officials: Uma M Borate, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu